CLINICAL TRIAL: NCT07013383
Title: The Effect of the "I Recycle, I Protect the Environment, I Leave a Livable World as a Legacy" Program on Recycling Behaviors of Secondary School Students
Brief Title: I Recycle, I Protect the Environment, I Leave a Livable World as a Legacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Feyza Bardak (Other)
Responsible Party: Sponsor-Investigator, Feyza Bardak, Suleyman Demirel University, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025/23
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Recycling; Behavior Change; Student
MeSH Terms: interventions — Recycling

STUDY DESIGN:
Masking Description: Masking will not be possible due to the method of application of this study. However, the data collector, statistician and reporting will be masked during the research process. In the research process, pre-test data will be collected by the teachers working in the study school. The post-test data will be collected by another researcher (a researcher trained in the data collection form and trained in the field of nursing student).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental)
  Interventions: Behavioral: "I Recycle, I Protect the Environment, I Leave a Livable World as a Legacy" Program

INTERVENTIONS:
Behavioral: "I Recycle, I Protect the Environment, I Leave a Livable World as a Legacy" Program — The training program includes topics such as environmental pollution, recycling behaviors, and the protection of natural resources and ecosystems. In addition, the program incorporates activities such as games, puzzle, brainstorming sessions, and the creation of painted cloth bags.
  Arms: Intervention Group

SUMMARY:
The research will be conducted to determine the effect of "I Recycle, I Protect the Environment, I Leave a Livable World as a Legacy" program on secondary school students' recycling behaviour.

DETAILED DESCRIPTION:
Recycling is crucial for environmental health as it plays a significant role in the protection of the environment, the conservation of natural resources, and the reduction of energy consumption. The Sustainable Development Goals (SDGs) are fundamentally centered around the themes of water management, energy sustainability, and responsible consumption and production practices. Without proactive measures to safeguard environmental health, the world is likely to encounter significant challenges related to water security, food supply, and the sustainability of natural resources in the future.

The study intervention was meticulously formulated on the basis of the Planned Behaviour Theory, encompassing a training programme focused on secondery school students' recycle behaviour. The training program includes topics such as environmental pollution, recycling behaviors, and the protection of natural resources and ecosystems. In addition, the program incorporates activities such as games, puzzle, brainstorming sessions, and the creation of painted cloth bags.

ELIGIBILITY:
Inclusion Criteria:

Being 10-14 years old and attend the school where the study is being conducted, Voluntarily agree to take part in the research,

Exclusion Criteria:

Having received previous education on environmental health

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Recycling Behavior Scale | T0 (Pre-test) T1 (15 days after the end of the procedure)
  Recycling Behavior Scale; The scale consists of a total of 14 items and three sub-dimensions. These sub-dimensions are stated as "participation" for the first factor, "valuation" for the second factor and "contribution to the economy" for the third factor. The scale explains 48.12% of the total variance. The total Cronbach alpha value of the scale is stated as 0.856.

SECONDARY OUTCOMES:
Recycling behavior predictive | T0 (Pre-test) T1 (15 days after the end of the procedure)
  The measure will be the number of implementations by students of 19 recycling behaviours predictive and defined on the basis of literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No